CLINICAL TRIAL: NCT02445456
Title: Feasibility of Sentinel Lymph Node Biopsy in Rectal Cancer
Acronym: SentiRect
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical difficulties in recruiting patients led to slower than expected recruitment. Recruitment was completely suspended during Covid and will not be restarted.
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Leeds (Other); Endomagnetics Ltd. (Industry)
Responsible Party: Principal Investigator, Chris Cunningham, Mr, Oxford University Hospitals NHS Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R37025/CN339
Record Dates: First submitted 2015-05-01; First posted 2015-05-15 (Estimated); Results first posted 2022-06-02 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Sentinel Lymph Node Biopsy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ex-vivo (Experimental): Patients with relatively advanced rectal cancer who are scheduled to undergo radical surgery to excise rectal tumour and mesorectum. They will receive endoscopic Sienna+ injection (magnetic tracer) 5 days before planned surgery. They will then undergo surgery to excise rectal cancer. The excised specimen will be examined using the Sentimag probe and by standard histology to assess for lymph nodes ex-vivo.
  Interventions: Drug: Sienna+ injection; Procedure: Surgery to excise rectal cancer; Device: Sentimag probe
- In-vivo (Experimental): Patients with early rectal cancer scheduled to undergo local excision of a rectal tumour by transanal endoscopic microsurgery (TEM). They will receive endoscopic Sienna+ injection (magnetic tracer) 5 days before planned surgery, and have an MRI scan to assess tracer spread. They will then undergo TEM surgery to excise the rectal cancer. During surgery the Sentimag probe will be used to locate the sentinel lymph node so it can be surgically removed. The excised specimen will be examined by standard histology.
  Interventions: Drug: Sienna+ injection; Other: MRI scan; Procedure: Surgery to excise rectal cancer; Device: Sentimag probe

INTERVENTIONS:
Drug: Sienna+ injection — Endoscopic injection of magnetic tracer
Other: MRI scan — MRI scan of pelvis to detect spread of magnetic tracer
  Arms: In-vivo
Procedure: Surgery to excise rectal cancer — Surgery as scheduled according to size and stage of rectal cancer. This will be either radical surgery or transanal endoscopic microsurgery (TEM)
Device: Sentimag probe — Probe to detect the previously injected magnetic tracer (Sienna+)

SUMMARY:
This study will assess whether the Sienna+/Sentimag system, which involves a magnetic tracer, is effective in identifying the sentinel lymph node in rectal cancer and whether it is then feasible to remove this lymph node during surgery to locally excise early rectal cancer.

DETAILED DESCRIPTION:
One issue in managing rectal cancer is identifying which patients will benefit from less radical surgery, which is much safer and better tolerated. However it does not remove lymph nodes where cancer cells may have spread. If lymph nodes containing cancer are left behind, the cancer may recur. So this surgery is only suitable in early rectal cancers not involving lymph nodes. Unfortunately, current investigations do not always accurately identify involved lymph nodes.

Sentinel lymph node biopsy (SLNB) is a technique to surgically remove the first lymph node where cancer cells spread. If this lymph node contains cancer, radical surgery is needed to reduce the risk of recurrence. However if it is clear, less radical surgery should be sufficient. This is standard practice for breast cancer and avoids unnecessary major surgery in many patients.

The investigators aim to assess whether SLNB is useful in rectal cancer. The investigators will determine whether the Sienna+/Sentimag system effectively identifies the sentinel lymph node, and whether the node can then be removed surgically.

The investigators will recruit patients in Oxford hospitals about to undergo surgery for rectal cancer. Patients will receive an injection of magnetic tracer during endoscopy prior to surgery. Some patients will have an extra MRI scan. During or after surgery, depending on the type of operation planned, a magnetic probe will be used to locate the sentinel lymph node in the tissue around the rectum. The removed specimen will be examined by a pathologist. Funding to undertake this study has been granted by the National Institute for Health Research (NIHR). Endomagnetics, the manufacturer, will supply the magnetic tracer and probe for use in this study.

If successful, the investigators will plan a larger clinical trial. This could have a major impact on improving outcomes for patients by allowing less radical surgery to be used where it is most appropriate.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with operable rectal cancer
* case discussed at Oxford Colorectal Cancer multi-disciplinary team (MDT) meeting
* willing and able to give informed consent
* willing and able to comply with all trial requirements, in the investigator's opinion

Exclusion Criteria:

* females who are pregnant or lactating
* known intolerance or hypersensitivity to iron, dextran compounds, magnetic tracers or superparamagnetic iron oxide particles (SPIO)
* cancer involvement of anal sphincter complex
* adults who are not able to give consent or are deemed vulnerable

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cunningham, MD FRCS, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ex-vivo: Patients with relatively advanced rectal cancer who are scheduled to undergo radical surgery to excise rectal tumour and mesorectum. They will receive endoscopic Sienna+ injection (magnetic tracer) 5 days before planned surgery. They will then undergo surgery to excise rectal cancer. The excised specimen will be examined using the Sentimag probe and by standard histology to assess for lymph nodes ex-vivo.
  Sienna+ injection: Endoscopic injection of magnetic tracer
  MRI scan: MRI scan of pelvis to detect spread of magnetic tracer
  Surgery to excise rectal cancer: Surgery as scheduled according to size and stage of rectal cancer. This will be either radical surgery or transanal endoscopic microsurgery (TEM)
  Sentimag probe: Probe to detect the previously injected magnetic tracer (Sienna+)
Period: Overall Study
Arm/Group | Ex-vivo | In-vivo
Started | 13 | 2
Completed | 13 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ex-vivo | In-vivo | Total
Number analyzed (Participants) | 13 | 2 | 15
Age, Customized [Count of Participants; unit: Participants]
  Age category: < 50 years | 2 | 1 | 3
  Age category: 51-60 years | 5 | 0 | 5
  Age category: 61-70 years | 6 | 0 | 6
  Age category: > 70 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 10 | 2 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 13 | 2 | 15
Pre-operative tumour T stage [Count of Participants; unit: Participants] — T component of the TNM (Tumour, Node, Metastasis) staging system, based on the pre-operative MRI scan.
  Participants
    mrT1 - tumour confined to inner bowel wall | 3 | 1 | 4
    mrT2 - tumour extending into muscle layer of the bowel wall | 5 | 1 | 6
    mrT3 - tumour has grown into the outer lining of the bowel wall | 5 | 0 | 5
Pre-operative N stage [Count of Participants; unit: Participants] — N component of the TNM (Tumour, Node, Metastasis) staging system, based on the pre-operative MRI scan.
  Participants
    mrN0 - no lymph nodes invaded by cancer cells | 10 | 2 | 12
    mrN1 - up to 3 nearby lymph nodes contain cancer cells | 2 | 0 | 2
    mrN2 - more than 3 lymph nodes contain cancer cells | 1 | 0 | 1
Prior treatment [Count of Participants; unit: Participants]
  Nil | 7 | 2 | 9
  Chemoradiation | 3 | 0 | 3
  Local excision | 3 | 0 | 3
Tumour diameter [Median (Full Range); unit: centimeter] | 3.0 [0.5 to 7.0] | 2.8 [2.0 to 3.5] | 3.0 [0.5 to 7.0]
Tumour height above anal margin [Median (Full Range); unit: centimeter] | 7 [1.5 to 15] | 11 [10 to 12] | 8 [1.5 to 15]
Tumour location [Count of Participants; unit: Participants]
  anterior | 4 | 1 | 5
  lateral | 4 | 0 | 4
  posterior | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing of Adverse or Hypersensitivity Reaction
Description: Assess frequency of any adverse of hypersensitivity reactions to tracer after endoscopic injection
Time Frame: 5 days after injection
Measure: Count of Participants; unit: Participants
Arm/Group | Ex-vivo | In-vivo
Number analyzed (Participants) | 13 | 2
Participants | 0 | 0

2. Primary Outcome: Number of Operations Where Effects of Tracer Injection Can be Detected by Surgeon During Surgery
Description: Assess frequency of Sienna+ tracer being detectable at the tumour injection site and in the lymph nodes at the time of surgery
Time Frame: at time of surgery
Population: Only patients who underwent surgery were analysed. Two patients in the ex-vivo group who were planned to have surgery did not proceed to surgery; instead they moved to a 'watch and wait' pathway after chemoradiation.
Measure: Number; unit: operations
Units Other Than Participants: Operations
Arm/Group | Ex-vivo | In-vivo
Number analyzed (Participants) | 11 | 2
Number analyzed (Operations) | 11 | 2
operations | 11 | 2

3. Primary Outcome: Number of Operations Where There Was Any Surgical Difficulty Due to Tracer Injection Based on Qualitative Assessment by Surgeon
Description: Surgeon's qualitative assessment of any difficulties encountered during surgery which could be attributable to prior injection of the tracer, such as pigmentation or fibrosis making surgery more difficult than normal
Time Frame: at time of surgery
Population: as for outcome 2
Measure: Number; unit: operations
Units Other Than Participants: Operations
Arm/Group | Ex-vivo | In-vivo
Number analyzed (Participants) | 11 | 2
Number analyzed (Operations) | 11 | 2
operations | 0 | 0

4. Secondary Outcome: Number of Mesorectal Specimens Which Demonstrated Correlation Between Histopathology and Sentimag Probe Findings for Lymph Node Number and Location
Description: The histopathology findings of lymph node distribution in the excised mesorectal specimen correlated with the information provided by the Sentimag probe.
Time Frame: 5 days after surgery
Population: Only patients who underwent radical surgery involving Total mesorectal excisison were included. The surgical specimens were analysed.
Measure: Number; unit: surgical mesorectal specimen
Units Other Than Participants: Surgical mesorectal specimens
Arm/Group | Ex-vivo | In-vivo
Number analyzed (Participants) | 11 | 1
Number analyzed (Surgical mesorectal specimens) | 11 | 1
surgical mesorectal specimen | 2 | 0

5. Secondary Outcome: Number of Mesorectal Specimens Which Demonstrated Coincidence Between Histopathological and Sentimag Probe Identification of the 'Sentinel' Lymph Node
Description: A pathologist will identify the sentinel lymph node histologically and record whether this matches the location identified by the Sentimag probe which has been previously marked with a suture
Time Frame: 5 days after surgery
Population: as for outcome 4
Measure: Number; unit: surgical mesorectal specimen
Units Other Than Participants: Surgical mesorectal specimens
Arm/Group | Ex-vivo | In-vivo
Number analyzed (Participants) | 11 | 1
Number analyzed (Surgical mesorectal specimens) | 11 | 1
surgical mesorectal specimen | 2 | 0

6. Secondary Outcome: High Resolution MRI Composite Map of Drainage Pattern of Sienna+ Tracer in Mesorectum
Description: Evaluation of individual variability in Sienna+ distribution after endoscopic injection on high resolution MRI scans to establish a baseline for individual variation
Time Frame: MRI scan done 2 hours after Sienna+ tracer injection
Population: Only patients who had MRI scans done following tracer injection were included.
Measure: Number; unit: MRI scans
Units Other Than Participants: MRI scans
Arm/Group | Ex-vivo | In-vivo
Number analyzed (Participants) | 9 | 2
Number analyzed (MRI scans) | 9 | 2
MRI scans
  tracer uptake by tumour | 6 | 1
  extraneous mucosal tracer uptake | 2 | 1
  tracer uptake by mesorectal nodes | 7 | 2
  Suspicious nodes on MRI after tracer injection | 3 | 1

7. Secondary Outcome: Number of TEM Operations Where the Sentinel Lymph Node Can be Identified and Removed
Description: Sentimag probe is used to localise the sentinel node during TEM (transanal endoscopic microsurgery) and then remove it if possible
Time Frame: at time of surgery
Population: This measure only applies to the In-vivo group. Ex-vivo group did not undergo TEM surgery.
Measure: Number; unit: TEM operations
Units Other Than Participants: TEM operations
Arm/Group | Ex-vivo | In-vivo
Number analyzed (Participants) | 0 | 1
Number analyzed (TEM operations) | 0 | 1
TEM operations |  | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the time between tracer injection until discharge from hospital after surgery. The range was 9-77 days due to differences in patient pathways.
Arm/Group | Ex-vivo | In-vivo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/2
Serious Adverse Events (participants affected / at risk) | 4/13 | 0/2
Other Adverse Events (participants affected / at risk) | 0/13 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ex-vivo (N=13) | In-vivo (N=2)
Post-operative ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anastomotic leak (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT02445456/Prot_SAP_000.pdf